CLINICAL TRIAL: NCT01295242
Title: Natural History of HPV Infections in Mid-Adult Women
Brief Title: Natural History of Human Papillomavirus (HPV) Infections in Mid-Adult Women (WHIM)
Acronym: WHIM
Status: Completed | Type: Observational
Sponsor: University of Washington (Other)
Responsible Party: Principal Investigator, Rachel Winer, Assistant Professor, University of Washington
Other Study IDs: 39810-C
Record Dates: First submitted 2011-02-02; First posted 2011-02-14 (Estimated); Last update posted 2013-11-19 (Estimated); Status verified 2013-11

CONDITIONS: Papillomavirus Infections
Keywords: HPV; Cervical Cancer
MeSH Terms: conditions — Papillomavirus Infections; Uterine Cervical Neoplasms

STUDY DESIGN:
Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Self-collected vaginal samples for HPV testing. Self-collected oral samples for HPV testing. Serum samples for HPV antibody testing.
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to determine rates of oral and genital human papillomavirus (HPV) infections, and look at risk factors for HPV infection in healthy mid-adult women.

DETAILED DESCRIPTION:
The investigators propose a longitudinal study of 500 women in order to determine rates and risk factors for HPV infections in 30-50 year old women. Participants will be followed for 6 months and will be asked to complete online questionnaires on their health, sexual behavior, HPV vaccinations, and cervical cancer screening. The investigators will ask participants to self-collect monthly vaginal swab samples and self-collect 2 oral swab samples. Women will also be asked to provide 2 blood samples. All swab samples will be tested for type-specific HPV deoxyribonucleic acid (DNA) using a polymerase chain reaction (PCR)-based assay, blood samples will be tested for HPV antibodies.

ELIGIBILITY:
Inclusion Criteria:

* affiliated with the University of Washington (student, staff, faculty)
* willing to self-collect vaginal samples at home for HPV testing
* able to provide informed consent

Exclusion Criteria:

* pregnant
* have had hysterectomy
* serious medical condition which prevents completion of activities of daily living

Ages: 30 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: 30 to 50 year old women affilitated with Univeristy of Washington (student, staff, faculty)
Sampling Method: Non-Probability Sample
Enrollment: 409 (Actual)
Dates: Start 2011-02; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Presence of type-specific HPV DNA in self-collected oral and vaginal swab samples | once a month for 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Rachel L Winer, PhD, MPH, Principal Investigator — University of Washington
Locations (1):
- University of Washington, Seattle, Washington, United States